CLINICAL TRIAL: NCT05066373
Title: A Phase 1, Single Centre, Open Label, Crossover Study in Healthy Volunteers Using Scintigraphy to Evaluate the Gastrointestinal Behaviour of EDP1815 Oral Dosage Forms.
Brief Title: Scintigraphy Study to Evaluate the Gastrointestinal Behavior of EDP1815 Oral Dosage Forms
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Evelo Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: EDP1815-104
Record Dates: First submitted 2021-09-23; First posted 2021-10-04 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Disintegration; Healthy
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EDP1815 capsule A (fasted) (Experimental): In part 1, 12 healthy volunteers will receive a single dose of EDP1815 capsule A, dosed in the fasted state
  Interventions: Drug: EDP1815 capsule A
- EDP1815 capsule B (fasted/fed) (Experimental): In part 1, 2 & 3, 12 healthy volunteers will receive a single dose of EDP1815 capsule B, dosed in the fasted and/or fed state
  Interventions: Drug: EDP1815 capsule B
- EDP1815 tablet (fasted/fed) (Experimental): In part 1, 3 & 4, 12 healthy volunteers will receive a single dose of EDP1815 tablet, dosed in the fasted and/or fed state
  Interventions: Drug: EDP1815 tablet

INTERVENTIONS:
Drug: EDP1815 capsule A — EDP1815 capsule A is an orally administered, pharmaceutical preparation of a single strain of Prevotella histicola. The capsule is radio-labeled with approximately 4 MBq 99mTc-DTPA
  Arms: EDP1815 capsule A (fasted)
Drug: EDP1815 capsule B — EDP1815 capsule B is an orally administered, pharmaceutical preparation of a single strain of Prevotella histicola. The capsule is radio-labeled with approximately 4 MBq 99mTc-DTPA
  Arms: EDP1815 capsule B (fasted/fed)
Drug: EDP1815 tablet — EDP1815 tablet is an orally administered, pharmaceutical preparation of a single strain of Prevotella histicola. The tablet is radio-labeled with approximately 4 MBq 99mTc-DTPA
  Arms: EDP1815 tablet (fasted/fed)

SUMMARY:
This study is to find out how different types of capsules or tablets containing EDP1815 move through the GI tract and release the drug after being swallowed. The capsules and tablets also contain a very small dose of a commonly used radioactive label called technetium-99m which is released in the GI tract to be seen on pictures taken by a scanner (gamma scintigraphy).

DETAILED DESCRIPTION:
This is a Phase I single centre, crossover, gamma scintigraphy study to investigate the gastrointestinal transit and disintegration kinetics of capsule and tablet formulations of EDP1815 (which contains a specific pure strain of Prevotella histicola, a natural human commensal organism).

In Part 1, up to 12 healthy male volunteers will receive single doses of EDP1815 administered either as capsules or tablets in 4 treatment periods.

The data generated in Part 1 will be assessed prior to progressing to Part 2 to select formulations and doses to be studied. Part 2 will include gamma scintigraphy in up to 12 healthy volunteers receiving single doses of EDP1815 capsules over up to 4 treatment periods.

The data generated in Part 2 will be assessed prior to progressing to Part 3 to select formulations and doses to be studied. Part 3 will include gamma scintigraphy in up to 12 healthy volunteers receiving single doses of EDP1815 capsules or tablets over up to 4 treatment periods.

The data generated in Part 3 will be assessed prior to progressing to Part 4 to select formulations and doses to be studied. Part 4 will include gamma scintigraphy in up to 12 healthy volunteers receiving single doses of EDP1815 tablets over up to 4 treatment periods.

Each capsule or tablet will contain the radio-isotope technetium-99m complexed to DTPA; 99mTc-DTPA, does not enter the systemic circulation and is routinely used for investigations of this type. Imaging via gamma scintigraphy will be used to assess the gut transit time and disintegration location/rate of the capsules/tablets. The drug will be given fasted or fed.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male
2. Body weight ≥50 kg and BMI 18-30 kg/m²
3. Healthy

Key Exclusion Criteria:

1. History or presence of any medical condition or abnormal laboratory test findings at screening that could affect the study conduct/results, or make the participant unlikely to fully complete the study or potentially adversely affect their safety due to taking part.
2. History of non-self-limiting gastrointestinal disorders, or currently suffering from disease known to impact gastric emptying, e.g. migraine, Type 1 or Type 2 diabetes mellitus.
3. Any contraindication to gamma scintigraphy.
4. Any non-removable metal objects such as metal plates, screws in the chest or abdominal area.
5. Total radiation dosimetry value which contraindicates participation.
6. Use of prescribed medication within 14 days prior to first dose which could interfere with the study procedures or affect gastric emptying and/or gut transit.
7. Use of over-the-counter (OTC) medication, including vitamins, pro and prebiotics and natural or herbal remedies, within 48 hours prior to first dose.
8. History of alcohol or other substance abuse.
9. Current smoker or recently discontinued smoking (less than 3 months).
10. History of allergy to any component of the dosage form or any other allergy which contraindicates participation.
11. Vegetarian or vegan.
12. Participation in this or another clinical study with an investigational drug within the prior 12 weeks, or more than four other clinical studies in the prior 12 month period.
13. Participants unwilling to comply with contraception requirements from first dose until 90 days (use of condom/spermicide in addition to use of protocol-specified highly effective contraception by female partners who could become pregnant)

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2021-08-09 (Actual); Primary Completion 2022-08-11 (Actual); Study Completion 2022-08-26 (Actual)

PRIMARY OUTCOMES:
Time to onset of radiolabel release | up to 12 hours
  The time to onset of disintegration/release for each EDP1815 formulation will be measured by using the time of onset of radiolabel release
Site of onset of radiolabel release | up to 12 hours
  The site of onset of disintegration/release for each EDP1815 formulation will be determined by using the site of onset of radiolabel release

SECONDARY OUTCOMES:
Gastric emptying time | up to 12 hours
  Gastrointestinal transit parameters will be measured using the gastric emptying time
Small intestinal transit time | up to 12 hours
  Gastrointestinal transit parameters will be measured using the small intestinal transit time
Colon arrival time | up to 12 hours
  Gastrointestinal transit parameters will be measured using the colon arrival time
Time to 50% release (T50) | up to 12 hours
  The radiolabel release kinetics of each EDP1815 formulation will be measured using the time to 50% release (T50)
Time to 90% release (T90) | up to 12 hours
  The radiolabel release kinetics of each EDP1815 formulation will be measured using the time to 90% release (T90)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Stevens, BPharm PhD, Principal Investigator — BDD Pharma Ltd
Locations (1):
- BDD Pharma Ltd, Glasgow, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No